CLINICAL TRIAL: NCT03472300
Title: Prevalence of Self-disclosed Knee Trouble and Use of Treatments Among Elderly Individuals From Frederiksberg Municipality - A Prospective Cohort Study
Brief Title: Prevalence of Self-disclosed Knee Trouble and Use of Treatments Among Elderly Individuals
Status: Active, not recruiting | Type: Observational
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Henning Bliddal, Head of the Parker Institute, Frederiksberg University Hospital
Other Study IDs: FrbCohort-01
Record Dates: First submitted 2018-03-13; First posted 2018-03-21 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis; Survey, Family Life; Complementary Therapies; Pain
Keywords: Knee Osteoarthritis; pain; Complementary Therapies; Survey; questionnaire
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Frederiksberg Citizens: All citizen in the Frederiksberg Community aged 60-69
  Interventions: Other: Survey about knee pain and treatment

INTERVENTIONS:
Other: Survey about knee pain and treatment — All citizens are surveyed to describe the prevalence of knee pain in a danish community.

SUMMARY:
Although knee pain is prevalent among community-dwelling older adults, little is known about how people in general handle their pain. We will conduct a survey to explore how knee pain affects people's lives and which treatments or self-management strategies they have chosen (or are being offered), and how these interact concerning pain reduction and maintenance of function.

DETAILED DESCRIPTION:
Although knee pain is prevalent among community-dwelling older adults and frequently leads to consultation in primary care, little is known about how people in general manage their knee pain.

Treatments of knee osteoarthritis include a variety of non-pharmaceutical, medical, and surgical interventions with highly individual and inconsistent results and with the possible exception of a longer lasting weight reduction, none of the non-surgical treatments have been able to demonstrate long-lasting effect on pain or disability.

It is well recognised that patient participation in handling of disease creates better compliance and satisfaction with pharmacological treatment.

Another option for taking active part in self-management is the use of complementary and alternative medicine (CAM). despite their popularity and effect, there is currently no overview of the actual extent of CAMs used for knee pain and disability at a population level, and most CAMs remain to be studied scientifically for efficacy.

The incidence of knee OA shows a steep increase at age above 60 years. Furthermore, after this age an increasing prevalence of disablement to knee trouble is encountered. To prevent this development, measures must be sought to alter the course of knee OA.

By asking people about how knee pain affects their life, which treatments or self-management strategies they have chosen (or are being offered), and how these interact for the reduction of pain and maintenance of function, new knowledge will be gained about the preferences and perceived effectiveness of treatments at large. The information gained will enable the prioritising of research on interventions to be tested and will align this with the primary concerns and interests of the population. This will subsequently lead to better guidance of patients by the health care providers, and will aid decision makers in choosing feasible health care policies and strategies.

ELIGIBILITY:
Inclusion Criteria:

* Between 60-69 years of age
* Citizen in the Community of Frederiksberg

Exclusion Criteria:

• No formal exclusion criteria but unability to understand/answer our questionnaire is per se an exclusion criteria

Ages: 60 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will comprise the sample of all elderly individuals 60-69 years old, living in the Frederiksberg municipality (central part of Copenhagen) Denmark
Sampling Method: Non-Probability Sample
Enrollment: 9600 (Estimated)
Dates: Start 2018-09-05 (Actual); Primary Completion 2028-10-21 (Estimated); Study Completion 2028-10-21 (Estimated)

PRIMARY OUTCOMES:
Self-disclosed knee trouble/pain | 1 Year
  Population incidence of self-disclosed knee trouble/pain

SECONDARY OUTCOMES:
Self-disclosed knee trouble/pain | Annually for 10 years
  Population incidence of self-disclosed knee trouble/pain
Knee injury and Osteoarthritis Outcome Score (KOOS) | Annually for 10 years
  Actual KOOS score and scores over time (respondents who report having knee pain)
Brief Illness Perception Questionnaire (IPQ-B) | Annually for 10 years
  Actual IPQ-B score and scores over time (respondents who report having knee pain). Generic questionnaire developed to measure illness perception. The IPQ-B contains eight items and one causal scale. Items 1-8 are rated using a 0-to-10 response scale, item 9 is a memo field. Five of the items assess cognitive illness representations: consequences (Item 1), timeline (Item 2), personal control (Item 3), treatment control (Item 4), and identity (Item 5). Two of the items assess emotional representations: concern (Item 6) and emotions (Item 8). One item assesses illness comprehensibility (Item 7).
  A low score on items number 1,2,5,6 and 8 indicates that the illness is perceived as benign while a low score on the items 3, 4 and 7 indicates that the illness is perceived as threatening. By reversing these three items it is possible to compute an overall score. A higher score reflects a more threatening view of the illness.
EQ-5D | Annually for 10 years
  Actual EQ-5D score and scores over time (all respondents)
Treatments of all kinds | Annually for 10 years
  To estimate the use of treatments of all kinds (both in the "established" health care system and as self-management), including use of non-pharmacological treatments
Influence of treatments (longitudinal) | Annually for 10 years
  Influence of treatments and their combination on use of health care system including surgical procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Ginnerup, Study Chair — The Parker Institute
Locations (1):
- the Parker Institute, Bispebjerg-Frederiksberg Hospital, Frederiksberg, Danmark, Denmark

REFERENCES:
- [Derived] Ginnerup-Nielsen E, Christensen R, Heitmann BL, Altman RD, March L, Woolf A, Bliddal H, Henriksen M. Prognostic value of illness perception on changes in knee pain among elderly individuals: Two-year results from the Frederiksberg Cohort study. Osteoarthr Cartil Open. 2023 Aug 19;5(4):100403. doi: 10.1016/j.ocarto.2023.100403. eCollection 2023 Dec. PMID 37671176
- [Derived] Ginnerup-Nielsen EM, Henriksen M, Christensen R, Heitmann BL, Altman R, March L, Woolf A, Karlsen H, Bliddal H. Prevalence of self-reported knee symptoms and management strategies among elderly individuals from Frederiksberg municipality: protocol for a prospective and pragmatic Danish cohort study. BMJ Open. 2019 Sep 4;9(9):e028087. doi: 10.1136/bmjopen-2018-028087. PMID 31488473